CLINICAL TRIAL: NCT00844090
Title: The Role of Apathy in Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLIN-011-08F
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Apathy; Diabetes
Keywords: Apathy; Diabetes; Self-care behaviors
MeSH Terms: conditions — Lethargy; Diabetes Mellitus | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Placebo Comparator): placebo tablets
  Interventions: Drug: methylphenidate or placebo
- Arm 2 (Experimental): methylphenidate tablets
  Interventions: Drug: methylphenidate or placebo

INTERVENTIONS:
Drug: methylphenidate or placebo — treat apathy to improve diabetes self care behaviors thereby improving glycemic control

SUMMARY:
In spite of several new medications and insulins for the control of blood sugars in patients with diabetes, a large number of patients do not have good control. This likely due to inability to carry out regular activities and self-care behaviors such as taking meds regularly, keeping a good diet, exercise etc. This inability to carry out self care lifestyle changes may be due to a condition called apathy. Apathy is a lack of motivation and persistence. In this study we will attempt to treat apathy with a medication called methylphenidate for 6 months and see if blood sugar/diabetes control improves.

DETAILED DESCRIPTION:
The incidence of diabetes in the US is at epidemic proportions. A large number of diabetes patients in the VA system have uncontrolled diabetes with high HbA1c. The inability to carry out important self-care behaviors such as measuring blood sugars regularly, following diet, exercise and medication programs may be due to apathy. Apathy is the lack of motivation, persistence and novelty. We have found this to be very prevalent in the VA diabetes population. We now do a randomized placebo controlled trial to see if treatment of apathy with methylphenidate will improve glycemic control in patients with A1c >8. Treatment will be for 6 months. The primary end point is HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Poor glycemic control HbA1c>8
* Presence of apathy, a score of >30 on AES
* Subjects should be on stable dose of metformin, thiozolidinediones, and sulfonylureas, statins and ACE inhibitors for at least two months
* Subjects should have a negative cardiac stress test within the previous year

Exclusion Criteria:

* Presence of major depressive disorder, psychosis, suicidal ideations, and history of stimulant dependence as evaluated by MINI.
* Patient currently being treated or a history hypersensitivity to methylphenidate
* Hypertension with BP>140/90
* History of renal disease with GFR<60
* History of hepatic failure with AST/ALT > three times the normal range
* History of seizure disorder, or Tourette's syndrome or presence of motor tics
* Patients with glaucoma
* Patients being treated with monoamine oxidase inhibitors (MAOIs) or Clonidine
* Patients with active cancer.
* Patients with acute illness needing hospitalization
* Patients with cardiovascular events such as myocardial infarction, stroke, amputation, unstable angina within the last six months.
* HbA1c> 12
* Planned elective surgery in next 6 months
* Pregnancy

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyrus DeSouza, MD, Principal Investigator — VA Medical Center, Omaha
Locations (1):
- VA Medical Center, Omaha, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period Oct 2009- Jan 2012.Participants recruited from Omaha VA outpatient clinics
Pre-assignment Details: All participants underwent a stress echo after consent. If stress echo was positive patient was not assigned to randomized arms
Groups:
- Methylphenidate: methylphenidate
  methylphenidate 10mg twice daily P.O. : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
- Placebo: placebo
  placebo only to treat apathy to improve diabetes self care behaviors thereby improving glycemic control
Period: Overall Study
Arm/Group | Methylphenidate | Placebo
Started | 52 | 54
Completed | 46 | 46
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Population: The number of participants for analysis was 92 in total since only 92 participants completed the study.
Groups:
- Methylphenidate: methylphenidate
  methylphenidate : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
- Placebo: placebo
  methylphenidate : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
- Total: Total of all reporting groups
Arm/Group | Methylphenidate | Placebo | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (9.9) | 56.0 (8.4) | 55.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 42 | 43 | 85

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Over Baseline
Description: measure of longer term glycemic control. A1c measured at baseline 6 weeks and 6 months
Time Frame: 6 months from baseline
Population: per protocol
Measure: Median (Standard Deviation); unit: percentage of HbA1c
Groups:
- Methylphenidate: methylphenidate
  methylphenidate 10mg BID P.O. : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
- Placebo: placebo
  Placebo tabs BID P.O. : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
Arm/Group | Methylphenidate | Placebo
Number analyzed (Participants) | 46 | 46
percentage of HbA1c | -1.0 (1.02) | -0.1 (1.04)

ADVERSE EVENTS:
Groups:
- Methyphenidate: methylphenidate
  methylphenidate 10mg bid p.o.: treat apathy to improve diabetes self care behaviors thereby improving glycemic control
- Placebo: placebo
  Placebo bid p.o. : treat apathy to improve diabetes self care behaviors thereby improving glycemic control
Arm/Group | Methyphenidate | Placebo
Serious Adverse Events (participants affected / at risk) | 7/46 | 6/46
Other Adverse Events (participants affected / at risk) | 28/46 | 25/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methyphenidate (N=46) | Placebo (N=46)
Blood Pressure and pulse (Cardiac disorders) | 2 (3) | 2 (2)
abdominal pain, nausea, loose stool (Gastrointestinal disorders) | 3 (3) | 2 (4) — adverse events only collected by organ system.
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
cellulitis (Infections and infestations) | 0 (0) | 1 (1) — hospitalization for cellulitis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methyphenidate (N=46) | Placebo (N=46)
gastrointestinal (Gastrointestinal disorders) | 20 (32) | 17 (24) — nausea , bloating collected as GI organ system.
fatigue (General disorders) | 5 (5) | 7 (7)
dizziness (General disorders) | 3 (3) | 1 (1) — mild self limited

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes